CLINICAL TRIAL: NCT00392886
Title: Dose Intensive Chemotherapy for Children Less Than Ten Years of Age Newly-Diagnosed With Malignant Brain Tumors: A Pilot Study of Two Alternative Intensive Induction Chemotherapy Regimens, Followed by Consolidation With Myeloablative Chemotherapy (Thiotepa and Carboplatin, With or Without Etoposide) and Autologous Stem Cell Rescue [HEAD START III]
Brief Title: Combination Chemotherapy With or Without Etoposide Followed By an Autologous Stem Cell Transplant in Treating Young Patients With Previously Untreated Malignant Brain Tumors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Jonathan L. Finlay, Childrens Hospital Los Angeles
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000503990; CHLA-HEAD-START-III; CHLA-HSIII; CHLA-2004-020; CHLA-04.020; UMN-MT2004-06
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2010-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood medulloblastoma; untreated childhood supratentorial primitive neuroectodermal tumor; childhood infratentorial ependymoma; childhood supratentorial ependymoma; newly diagnosed childhood ependymoma; childhood high-grade cerebral astrocytoma; childhood oligodendroglioma; childhood atypical teratoid/rhabdoid tumor; childhood choroid plexus tumor; untreated childhood cerebellar astrocytoma; untreated childhood visual pathway and hypothalamic glioma; untreated childhood pineoblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Rhabdoid Tumor; Choroid Plexus Neoplasms | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; Methotrexate; Temozolomide; Thiotepa; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

ARMS (2):
- Regimen C (Experimental): Patients receive induction therapy of vincristine IV on days 1, 8, and 15 of courses 1-3, oral temozolomide once daily on days 1-5, and carboplatin IV over 4 hours on days 1 and 2. Patients also receive G-CSF SC beginning on day 6 and continuing until blood counts recover. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients receive consolidation therapy of carboplatin IV over 4 hours on days -8 to -6 and thiotepa IV over 3 hours on days -5 to -3, undergo reinfusion of bone marrow or peripheral blood stem cells on day 0, and receive G-CSF SC beginning on day 1 and continuing until blood counts recover. Beginning within 6 weeks after transplantation, some patients undergo radiotherapy once daily 5 days a week for 4-6 weeks in the absence of disease progression or unacceptable toxicity and some patients undergo radiotherapy if there is evidence of tumor remaining after completion of induction chemotherapy.
  Interventions: Drug: carboplatin; Drug: temozolomide; Drug: thiotepa; Drug: vincristine sulfate; Procedure: autologous bone marrow transplantation; Procedure: autologous hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy
- Regimen D2 (Experimental): In courses 1, 3, and 5, patients receive cisplatin IV over 6 hours on day 1, cyclophosphamide IV over 1 hour and etoposide IV over 2 hours on days 2 and 3, high-dose methotrexate IV over 4 hours on day 4, vincristine IV on days 1, 8, and 15 (in courses1 and 3), and filgrastim (G-CSF) subcutaneously (SC) beginning on day 5 and continuing until blood counts recover. In courses 2 and 4, patients receive oral temozolomide once daily on days 1-5, oral etoposide once daily on days 1-10, cyclophosphamide IV over 1 hour on days 11 and 12, vincristine IV on days 1, 8, and 15 (in course 2), and G-CSF SC beginning on day 13 and continuing until blood counts recover. Patients receive consolidation therapy as in regimen C in combination with etoposide IV over 3 hours on days -5 to -3 and undergo autologous bone marrow or peripheral blood stem cell transplantation, receive G-CSF, and undergo radiotherapy as in regimen C.
  Interventions: Drug: carboplatin; Drug: cisplatin; Drug: cyclophosphamide; Drug: etoposide; Drug: methotrexate; Drug: temozolomide; Drug: thiotepa; Drug: vincristine sulfate; Procedure: autologous bone marrow transplantation; Procedure: autologous hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin — Given IV
Drug: cisplatin — Given IV
  Arms: Regimen D2
Drug: cyclophosphamide — Given IV
  Arms: Regimen D2
Drug: etoposide — Given IV and orally
  Arms: Regimen D2
Drug: methotrexate — Given IV
  Arms: Regimen D2
Drug: temozolomide — Given orally
Drug: thiotepa — Given IV
Drug: vincristine sulfate — Given IV
Procedure: autologous bone marrow transplantation — Given on day 0
Procedure: autologous hematopoietic stem cell transplantation — Given on day 0
Procedure: peripheral blood stem cell transplantation — Given on day 0
Radiation: radiation therapy — Some patients undergo radiation therapy once daily, 5 days a week for 4-6 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. A bone marrow or peripheral stem cell transplant using stem cells from the patient may be able to replace blood-forming cells that were destroyed by chemotherapy. This may allow more chemotherapy to be given so that more tumor cells are killed.

PURPOSE: This phase III trial is studying how well giving combination chemotherapy with or without etoposide followed by an autologous stem cell transplant works in treating young patients with previously untreated malignant brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 2-year event-free survival (EFS) and overall survival (OS) of pediatric patients with previously untreated nondisseminated medulloblastoma (< 4 years of age), disseminated medulloblastoma (< 10 years of age), or noncerebellar primitive neuroectodermal tumors (PNET) (disseminated or non-disseminated) treated with induction chemotherapy followed by consolidation with myeloablative chemotherapy and autologous hematopoietic stem cell rescue.
* Determine the toxicity of this regimen in these patients.
* Determine the mortality of patients treated with this regimen.

Secondary

* Determine the complete and partial response rates after completion of induction chemotherapy in these patients stratified according to pathology (medulloblastoma vs noncerebellar PNET vs high-grade gliomas vs atypical teratoid/rhabdoid tumors vs choroid plexus carcinomas and atypical papillomas vs ependymomas).
* Describe the EFS and OS of these patients stratified according to additional diagnoses (atypical teratoid/rhabdoid tumors vs choroid plexus carcinomas and atypical choroid plexus papillomas vs ependymomas vs high-grade gliomas).
* Describe the time to progression and patterns of relapse in these patients stratified by diagnosis and radiotherapy received (< 6 years of age with evidence of no residual tumor pre-transplant and no post-transplant consolidation radiotherapy vs < 6 years of age with residual tumor present pre-transplant treated with post-transplant consolidation radiotherapy vs > 6 years of age treated with post-transplant consolidation radiotherapy).
* Determine the neuropsychometric function, endocrinologic function, and physical growth in these patients stratified according to radiotherapy received (none vs reduced-volume craniospinal radiotherapy vs focused local-field radiotherapy).

OUTLINE: This is a pilot study. Patients are stratified according to type of tumor (nonglial vs glial and diffuse pontine).

* Regimen C (patients with glial tumors):

  * Stem cell harvesting (bone marrow and/or peripheral blood): Patients undergo leukapheresis or bone marrow aspiration to collect bone marrow or peripheral blood stem cells prior to beginning induction chemotherapy or after the first course of induction chemotherapy.
  * Induction chemotherapy: Patients receive vincristine IV on days 1, 8, and 15 of courses 1-3, oral temozolomide once daily on days 1-5, and carboplatin IV over 4 hours on days 1 and 2. Patients also receive G-CSF SC beginning on day 6 and continuing until blood counts recover. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients with unresectable bulky disease and corticosteroid dependence are removed from study. All other patients proceed to consolidation chemotherapy.

* Consolidation chemotherapy: Patients receive carboplatin IV over 4 hours on days -8 to -6 and thiotepa IV over 3 hours on days -5 to -3.
* Autologous bone marrow or peripheral blood stem cell transplantation: Patients undergo reinfusion of bone marrow or peripheral blood stem cells on day 0. Patients also receive G-CSF SC beginning on day 1 and continuing until blood counts recover.
* Radiotherapy: Beginning within 6 weeks after stem cell transplantation, patients > 6 years of age at diagnosis undergo radiotherapy once daily 5 days a week for 4-6 weeks in the absence of disease progression or unacceptable toxicity. Patients ≤ 6 years of age undergo radiotherapy if there is evidence of tumor remaining after completion of induction chemotherapy.

  * Regimen D2 (patients with nonglial tumors):
* Stem cell harvesting (bone marrow and/or peripheral blood): Patients undergo leukapheresis or bone marrow aspiration to collect bone marrow or peripheral blood stem cells prior to beginning induction chemotherapy or after the first course of induction chemotherapy.
* Induction chemotherapy:

  * Courses 1, 3, and 5 (28 days per course): Patients receive cisplatin IV over 6 hours on day 1, cyclophosphamide IV over 1 hour and etoposide IV over 2 hours on days 2 and 3, high-dose methotrexate IV over 4 hours on day 4, and filgrastim (G-CSF) subcutaneously (SC) beginning on day 5 and continuing until blood counts recover. Patients also receive vincristine IV on days 1, 8, and 15 of courses 1 and 3.
  * Courses 2 and 4 (28 days per course): Patients receive oral temozolomide once daily on days 1-5, oral etoposide once daily on days 1-10, cyclophosphamide IV over 1 hour on days 11 and 12, and G-CSF SC beginning on day 13 and continuing until blood counts recover. Patients also receive vincristine IV on days 1, 8, and 15 of course 2.

Patients with unresectable bulky disease and corticosteroid dependence are removed from study. All other patients proceed to consolidation chemotherapy.

* Consolidation chemotherapy: Patients receive carboplatin IV over 4 hours on days -8 to -6 and thiotepa IV over 3 hours and etoposide IV over 3 hours on days -5 to -3.
* Autologous bone marrow or peripheral blood stem cell transplantation: Patients undergo re-infusion of bone marrow or peripheral blood stem cells on day 0. Patients also receive G-CSF SC beginning on day 1 and continuing until blood counts recover.
* Radiotherapy:Patients undergo radiotherapy as in regimen C. Patients in both regimens undergo neuropsychological testing after induction chemotherapy but before consolidation chemotherapy and then at 18, 36, and 54 months after completion of study treatment. Neuropsychometric and neuroendocrine testing is performed before and after radiotherapy. Quality of life is also assessed periodically.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant brain tumor, including any of the following:

  * Posterior fossa medulloblastoma/primitive neuroectodermal tumor (PNET)*

    * All stages allowed
    * Must be < 4 years of age at diagnosis unless there is evidence of postoperative residual tumor (> 1.5 cm² tumor area) or evidence of neuraxis or extraneural dissemination (high-stage)
    * Medulloblastoma, cerebral neuroblastoma, and ependymoblastoma allowed

      * Low-stage (standard-risk) medulloblastoma not allowed in patients > 4 years of age
  * Ependymoma*

    * All stages and locations allowed
    * Cellular and anaplastic subtypes allowed (no myxopapillary ependymomas of the spinal cord)
    * Must be < 36 months of age at diagnosis for posterior fossa tumor OR < 72 months of age for supratentorial tumor
    * Evidence of neuraxis dissemination irrespective of primary site
    * No cellular (low-grade) supratentorial ependymomas at any age with complete resection of parenchymally based (i.e., not periventricular) supratentorial tumors
  * Brain stem tumor*

    * All stages allowed irrespective of extent of resection
    * No unbiopsied diffuse intrinsic pontine tumor
    * Tumor pathologically confirmed to be either malignant glioma or PNET allowed
  * High-grade glioma**
  * Primary atypical teratoid/rhabdoid tumor of the CNS*
  * Choroid plexus carcinoma or atypical choroid plexus papilloma*

    * All stages and locations allowed
  * Anaplastic astrocytoma**
  * Glioblastoma multiforme**
  * Anaplastic oligodendroglioma**
  * Anaplastic ganglioglioma**
  * Other anaplastic mixed gliomas**
  * Small-cell glioblastoma**
  * Giant-cell glioblastoma**
  * Gliosarcoma**
* The following diagnoses or subtypes are not allowed:

  * Choroid plexus papilloma
  * Pineocytoma
  * Low-grade mixed glioma
  * Primary CNS germ cell tumor
  * Primary CNS lymphoma
  * Solid leukemic lesions (i.e., chloromas, granulocytic sarcomas)
  * Pleomorphic xanthoastrocytoma, low grade
  * Desmoplastic ganglioglioma
  * Low-grade astrocytoma
* Previously untreated disease
* Has undergone definitive surgery within the past 42 days NOTE: *Patients receive treatment according to regimen D2

NOTE: **Patients receive treatment according to regimen C

PATIENT CHARACTERISTICS:

* Bilirubin < 1.5 mg/dL
* ALT and AST < 2.5 times upper limit of normal
* Creatinine clearance and/or glomerular filtration rate ≥ 60 mL/min

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy or chemotherapy
* Prior corticosteroids allowed
* No concurrent corticosteroids for antiemesis only
* No concurrent brachytherapy or electron radiotherapy
* No concurrent dairy products or grapefruit juice with temozolomide administration

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2004-03; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Time to tumor progression, disease recurrence, or death of any cause
Event-free survival at 2 years
Toxicity

SECONDARY OUTCOMES:
Response to induction as assessed by one-time tumor measurements at baseline and after completion of induction chemotherapy
Time to death
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan L. Finlay, MB, ChB, Study Chair — Children's Hospital Los Angeles; Girish Dhall, MD — Children's Hospital Los Angeles; Kelley Haley, RN, BSN — Children's Hospital Los Angeles
Locations (37):
- United States (29):
  - Phoenix Children's Hospital Outpatient Center, Phoenix, Arizona
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Clinic, Jacksonville, Florida
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Riley's Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Tomorrows Children's Institute at Hackensack University Medical Center, Hackensack, New Jersey
  - Schneider Children's Hospital, New Hyde Park, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (3):
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Hospital for Sick Children, Toronto, Ontario
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - Wellington Children's Hospital, Wellington
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Universitaets Kinderklinik, Bern